CLINICAL TRIAL: NCT02190968
Title: Reducing Residual Depressive Symptoms With Web-based Mindful Mood Balance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: University of Colorado, Boulder (Other); Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Zindel Segal, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH102229-01A1 (NIH)
Record Dates: First submitted 2014-07-10; First posted 2014-07-15 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Major Depressive Disorder, Recurrent, in Remission; Depressive Symptoms
Keywords: Mindfulness Based Cognitive Therapy; Internet interventions; Residual depressive symptoms; Depressive relapse prevention
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Mood Balance (Experimental): An 8 session internet intervention targeting residual depressive symptoms.
  Interventions: Behavioral: Usual Depression Care; Behavioral: Mindful Mood Balance
- Usual Depression Care (Active Comparator): Usual Depression Care through Kaiser Permanente Colorado
  Interventions: Behavioral: Usual Depression Care

INTERVENTIONS:
Behavioral: Usual Depression Care — Usual Depression Care will be based on the Kaiser Permanente Adult Depression National Guidelines - an adaptation of STAR*D (Rush et al., 2006) for antidepressant management and the IMPACT (Unitzer et al., 2002; 2008) model for therapy.
Behavioral: Mindful Mood Balance — Mindful Mood Balance is an individually tailored, web-based version of Mindfulness-Based Cognitive Therapy, a manualized, group skills training program (Segal et al., 2002) that is based on an integration of aspects of cognitive therapy for depression (Beck, 1979) with components of the mindfulness-based stress reduction program (Kabat-Zinn, 1990). Patients participated in 8 internet sessions, each of which incorporates didactic and experiential learning, along with home practice of skills taught in the program.
  Arms: Mindful Mood Balance

SUMMARY:
Many patients report residual depressive symptoms despite seemingly successful treatment. With the investigators' previous funding, we developed - Mindful Mood Balance - an online treatment that targets RDS by teaching specific emotion regulation and depression self-management skills that are entirely compatible with antidepressant treatment. The investigators now propose a controlled study to determine whether MMB is more effective than usual care at reducing RDS and other key outcomes. If successful, MMB's online delivery format would provide high fidelity and low-cost empirically supported management of residual symptoms, leading to more robust remission, improved functioning and sustained recovery from MDD over time.

DETAILED DESCRIPTION:
Residual depressive symptoms (RDS) following remission of major depressive disorder (MDD) are reported by 80-90% of adults receiving first-line antidepressant pharmacotherapy and carry an elevated risk for a chronic course of illness, rapid relapse and functional impairment. Strategies for managing residual symptoms, however, have met with mixed success. Mindful Mood Balance (MMB; R34 MH0877223) is an individually tailored, web-based treatment designed to train remitted depressed patients to disengage from dysphoria-activated depressogenic thinking that perpetuates RDS and increases risk for relapse/recurrence. MMB was developed to increase access to Mindfulness-Based Cognitive Therapy (MBCT; R01 MH066992), an empirically supported prophylactic group treatment that can be easily sequenced with acute phase antidepressant pharmacotherapy. Results from our open trial of MMB (N=100) showed an effect size of d=1.09 for pre to post treatment reductions in depression scores among patients with RDS and d=1.54 in a quasi-experimental comparison to patients receiving usual care, with an on average reduction of 1.98 points on the PHQ-9 for MMB patients. The investigators now propose a pragmatic randomized clinical trial of MMB to evaluate its effectiveness in reducing RDS in recurrently depressed patients. Patients will be members of Kaiser-Permanente Colorado (N = 460), aged 18 to 75, who score >5 and <9 on the PHQ-9, in remission from MDD and will be randomized 1:1 to either the usual depression care pathway (DepCare) or Mindful Mood Balance (MMB)+DepCare.

The investigators plan to test whether patients receiving MMB+DepCare will show greater reductions in RDS at both 8 week and 12 months follow up, than those receiving DepCare alone. The investigators are also interested in examining whether fewer patients in MMB+DepCare will relapse over the follow up and will have higher end state functioning and quality of life. In order to examine the costs associated with adding this online treatment to the Depression Care Pathways at KPCO, the investigators will calculate the marginal costs per additional number of depression free days (DFDs) for patients. Resolution of RDS can reduce the enormous personal and social costs experienced by Americans with this persistent symptom burden.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a PHQ-9 score between 5 and 9
* At least one prior episode of MDD

Exclusion Criteria:

* presence of schizophrenia or current psychosis, organic mental disorder or pervasive developmental delay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 | Change from Baseline to 12 weeks and 15 months
  Changes in self reported depressive symptom severity
Patient Health Questionnaire-9 | Between 12 weeks and 15 months
  Rates of depressive relapse, defined as patients who score 15 or greater on the PHQ-9
Patient Health Questionnaire-9 | Between baseline to 12 weeks.
  Conversion from moderate/high risk to low risk symptom categories, defined as a patient whose PHQ-9 score drops from a baseline PHQ-9 score between 5 and 9 to a mean score of 4 or less

SECONDARY OUTCOMES:
Ruminative Responses Scale | Change from Baseline to 6 weeks, 12 weeks and 15 months
  A self-report measure of rumination
Five Facet Mindfulness Questionnaire | Change from Baseline to 6 weeks, 12 weeks and 15 months
  Self report measure of mindful awareness
Five Facet Mindfulness Scale | Change from Baseline to 6 weeks, 12 weeks and 15 months
  Self report measure of mindful awareness
Experiences Questionnaire | Change from Baseline to 6 weeks, 12 weeks and 15 months
  Self report measure of decentering/wider awareness

OTHER OUTCOMES:
Depression Free Days | Change from Baseline to 12 weeks and 15 months
  Self report of days free of depression
Generalized Anxiety Disorder Assessment - 7 | Change from Baseline to 12 weeks and 15 months
  Self report measure of generalized anxiety
Short Form Health Survey - 12 | Change from Baseline to 12 weeks and 15 months
  Self report measure of physical and mental health
Emotion Dot Probe Task | Change from Baseline to 12 weeks and 15 months
  A behavioural measure of attentional bias

CONTACTS AND LOCATIONS:
Overall Officials: Zindel V Segal, PhD, Principal Investigator — University of Toronto
Locations (1):
- Kaiser Permanente Institute for Health Research, Denver, Colorado, United States

REFERENCES:
- [Background] Boggs JM, Beck A, Felder JN, Dimidjian S, Metcalf CA, Segal ZV. Web-based intervention in mindfulness meditation for reducing residual depressive symptoms and relapse prophylaxis: a qualitative study. J Med Internet Res. 2014 Mar 24;16(3):e87. doi: 10.2196/jmir.3129. PMID 24662625
- [Background] Segal ZV, Bieling P, Young T, MacQueen G, Cooke R, Martin L, Bloch R, Levitan RD. Antidepressant monotherapy vs sequential pharmacotherapy and mindfulness-based cognitive therapy, or placebo, for relapse prophylaxis in recurrent depression. Arch Gen Psychiatry. 2010 Dec;67(12):1256-64. doi: 10.1001/archgenpsychiatry.2010.168. PMID 21135325
- [Background] Dimidjian S, Beck A, Felder JN, Boggs JM, Gallop R, Segal ZV. Web-based Mindfulness-based Cognitive Therapy for reducing residual depressive symptoms: An open trial and quasi-experimental comparison to propensity score matched controls. Behav Res Ther. 2014 Dec;63:83-9. doi: 10.1016/j.brat.2014.09.004. Epub 2014 Sep 18. PMID 25461782
- [Derived] Boggs JM, Ritzwoller DP, Beck A, Dimidjian S, Segal ZV. Cost-Effectiveness of a Web-Based Program for Residual Depressive Symptoms: Mindful Mood Balance. Psychiatr Serv. 2022 Feb 1;73(2):158-164. doi: 10.1176/appi.ps.202000419. Epub 2021 Jul 29. PMID 34320822
- [Derived] Segal ZV, Dimidjian S, Beck A, Boggs JM, Vanderkruik R, Metcalf CA, Gallop R, Felder JN, Levy J. Outcomes of Online Mindfulness-Based Cognitive Therapy for Patients With Residual Depressive Symptoms: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Jun 1;77(6):563-573. doi: 10.1001/jamapsychiatry.2019.4693. PMID 31995132
- See also: Mindfulness Based Cognitive Therapy Website — http://mbct.com/